CLINICAL TRIAL: NCT00005048
Title: Safety and Efficacy of One Hour Weekly Taxol Infusion and Estramustine in Hormone Refractory Prostate Cancer
Brief Title: Estramustine and Paclitaxel in Treating Patients With Prostate Cancer That Has Not Responded to Hormone Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000067640; NYU-9715; NCI-G00-1716
Record Dates: First submitted 2000-04-06; First posted 2004-06-18 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2000-11

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Estramustine; Paclitaxel

INTERVENTIONS:
Drug: estramustine phosphate sodium
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining estramustine and paclitaxel in treating patients who have prostate cancer that has not responded to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose (MTD) of paclitaxel with estramustine in patients with hormone refractory prostate cancer. II. Evaluate the toxicity of this combination at the MTD of paclitaxel in this patient population. III. Determine any objective tumor response arising from this treatment in these patients.

OUTLINE: This is a dose escalation study of paclitaxel. Patients receive oral estramustine daily on days 1-3 and paclitaxel IV over 1 hour on day 3 weekly for 6 weeks followed by 1 week of rest. Treatment continues for at least 2 courses in the absence of unacceptable toxicity or disease progression. Cohorts of 3-6 patients receive escalating doses of paclitaxel until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicities.

PROJECTED ACCRUAL: A minimum of 18 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed adenocarcinoma of the prostate with progressive systemic disease despite at least 1 endocrine manipulation including 1 of the following: Orchiectomy LHRH analogue with or without flutamide, megestrol, or diethylstilbestrol Flutamide must be discontinued for at least 2 weeks with PSA stabilized above normal or rising Measurable or evaluable disease No brain metastasis

PATIENT CHARACTERISTICS: Age: Not specified Performance status: ECOG 0-2 Life expectancy: Greater than 2 months Hematopoietic: Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin greater than 1 mg/dL SGOT greater than 2 times upper limit of normal Renal: Creatinine less than 2 mg/dL Hydronephrosis with impaired renal function must be decompressed adequately Cardiovascular: No severe cardiac (i.e., symptomatic arrhythmia requiring medication or active congestive heart failure) or coronary disease that are unstable despite medication Other: Adequate nutritional status (at least 1,500 Kcal/day) No other significant active medical illness that would preclude study therapy or survival No other malignancy within the past 5 years except adequately treated basal or squamous cell carcinoma of the skin No acute spinal cord compression

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent biologic response modifiers Chemotherapy: No other concurrent chemotherapy Endocrine therapy: See Disease Characteristics At least 2 weeks since prior corticosteroids No concurrent exogenous corticosteroids except for documented CNS metastases or adrenal insufficiency Concurrent hormones for nondisease conditions allowed (e.g., insulin for diabetes mellitus) Concurrent continuation of monthly hormonal therapy with an LHRH agonist or DES required Radiotherapy: Prior radiation to symptomatic metastatic site allowed provided it is not the only measurable or evaluable lesion At least 2 weeks since prior radiotherapy and recovered No concurrent radiotherapy No concurrent palliative radiotherapy except for whole brain irradiation for documented CNS disease or impending spinal cord compression Surgery: See Disease Characteristics At least 3 weeks since prior surgery and recovered Other: No other concurrent treatment for prostate cancer except pain palliation

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1997-04; Primary Completion 2000-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Chachoua, MD, Study Chair — NYU Langone Health
Locations (2):
- United States (2):
  - Kaplan Cancer Center, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York